CLINICAL TRIAL: NCT04682145
Title: Adverse Event Data Collection From the EUHASS Registry on Turoctocog Alfa Pegol
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7088-4557; U1111-1235-5939 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Haemophilia A patients: All patients with haemophilia A treated with turoctocog alfa pegol and reporting adverse events to EUHASS.
  Interventions: Drug: Turoctocog alfa pegol

INTERVENTIONS:
Drug: Turoctocog alfa pegol — Patients will be treated with commercially available turoctocog alfa pegol according to routine clinical practice at the discretion of the treating physician. A decision to initiate treatment with commercially available turoctocog alfa pegol has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in the registry in scope.

SUMMARY:
This non-interventional study concerns a safety data collection based on adverse event data from a third-party registry (European Haemophilia Safety Surveillance System, EUHASS) that includes information about adverse events from patients with haemophilia A treated with turoctocog alfa pegol. There is no extra burden to the patients by participating in this registry-based data collection.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the European Haemophilia Safety Surveillance System (EUHASS).

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with haemophilia A treated with turoctocog alfa pegol and reporting adverse events to EUHASS.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) reported to the registry with suspected relation to turoctocog alfa pegol, Adverse Drug Reactions (ADRs), in patients with haemophilia A for renal, hepatic and neurological events. | From start to end of data collection (December 2019 to January 2025)
  Count

SECONDARY OUTCOMES:
Other AEs reported to the registry during the study period with suspected relation to turoctocog alfa pegol in patients with haemophilia A | From start to end of data collection (December 2019 to January 2025)
  Count. Includes ADRs of special interest (de novo FVIII inhibitors equal to or above 0.6 Bethesda Units (BU)); anaphylaxis and other allergic reactions; thromboembolic events).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor & Disclosure (2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Søborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com